CLINICAL TRIAL: NCT06282757
Title: The Effect of Physiotherapists' Placebo or Nocebo Communication About Virtual Reality on Treatment Beliefs in Patients With CMP
Brief Title: Physiotherapists' Placebo or Nocebo Communication Regarding VR in CMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HAN University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Bart Staal, Professor (lector), HAN University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 202302
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Communication; Chronic Pain
MeSH Terms: conditions — Communication; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Experimental): The placebo intervention group will be shown an online educational VR video.
  Interventions: Other: Video placebo communication
- Nocebo group (Active Comparator): The nocebo intervention group will be shown an online educational VR video.
  Interventions: Other: Video nocebo communication

INTERVENTIONS:
Other: Video placebo communication — The placebo communication video comprises of an educational VR video containing placebo enhancing verbal language.
  Arms: Placebo group
Other: Video nocebo communication — The nocebo communication video comprises of an educational VR video containing nocebo stimulating verbal language.
  Arms: Nocebo group

SUMMARY:
Rationale: Chronic musculoskeletal pain (CMP) is a common and disabling condition. Physiotherapy is the most frequently administered non-pharmacological treatment option for patients with CMP and recently virtual reality (VR) was introduced in physiotherapy care as a novel treatment modality. Proper communication about physiotherapy treatment (modalities) is important to improve treatment outcomes, by applying placebo effects enhancing communication and avoiding nocebo effects enhancing communication. However, yet is still unknown to what extent this applies to communication of physiotherapists about VR in patients with CMP.

Objective: To determine the effect of physiotherapists' placebo or nocebo therapeutic communication about VR, on treatment credibility and expectation in patients with CMP

Study design: Web-based randomized controlled trial.

Study population: 100 participants

Intervention: The placebo intervention group will be shown an educational video about VR, containing placebo effects enhancing verbal language. The nocebo intervention group will be shown an educational video about VR, containing nocebo effects enhancing verbal language.

Primary study parameters: The primary study parameters are treatment credibility and treatment expectation. Treatment credibility and treatment expectations will be measured using the Dutch credibility and expectancy questionnaire (CEQ).

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18
* access to the internet
* provide informed consent
* suffers from CMP

Exclusion Criteria:

* lacked comprehension of the Dutch language
* had experience with therapeutic VR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in treatment expectancy measured using the Credibility and Expectancy Questionnaire (CEQ) | Baseline and immediately after the intervention
  This questionnaire on treatment expectancy scores from 6 (lowest expectancy) to 54 (highest expectancy)
Change in treatment credibility measured using the Credibility and Expectancy Questionnaire (CEQ) | Baseline and immediately after the intervention
  This questionnaire on treatment credibility scores from 5 (lowest credibility) to 45 (highest credibility)

SECONDARY OUTCOMES:
Change in openness to VR measured using a single question | Baseline and immediately after the intervention
  The question "would you be open to treatment with therapeutic VR" was scored with a yes/no
Change in pain intensity measured using the Numeric Pain Rating Scale (NPRS) | Baseline and immediately after the intervention
  This questionnaire on pain intensity scores from 0 (no pain) to 10 (maximal pain)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Staal, PhD, Principal Investigator — HAN University of Applied Sciences
Locations (1):
- HAN University of Applied Sciences, Nijmegen, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No
Not planned to share IPD